CLINICAL TRIAL: NCT05442983
Title: A Randomized, Single-center, Single-blind, Placebo-controlled Study to Evaluate the Efficacy of PanCytoVir™ 500 mg Twice Daily and 1000 mg Twice Daily for the Treatment of Non-hospitalized Patients With COVID-19 Infection
Brief Title: A Study to Evaluate the Efficacy of PanCytoVir™ for the Treatment of Non-Hospitalized Patients With COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TrippBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID-19/01/05/2022
Record Dates: First submitted 2022-06-30; First posted 2022-07-05 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Probenecid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PanCytoVir™ 500 mg twice daily (Experimental)
  Interventions: Drug: PanCytoVir™ (probenecid)
- PanCytoVir™ 1000 mg twice daily (Experimental)
  Interventions: Drug: PanCytoVir™ (probenecid)
- Placebo twice daily (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PanCytoVir™ (probenecid) — Active drug
  Arms: PanCytoVir™ 1000 mg twice daily; PanCytoVir™ 500 mg twice daily
Drug: Placebo — Matching placebo
  Arms: Placebo twice daily

SUMMARY:
This is a randomized, single-center, single-blind, placebo controlled, study to evaluate efficacy of PanCytoVir™ 500 mg twice daily and 1000 mg twice daily for the treatment of non-hospitalized patients with COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Non-hospitalized Patients with RT-PCR confirmed COVID-19 in ≤ 48 hours prior to randomization.
2. Patients with WHO Ordinal Scale score 1 and 2.
3. Patient has presented within 5 days or less of randomization with at least one early onset COVID-19 symptom (i.e. fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, vomiting or diarrhea).
4. Men and non-pregnant women, 18 - 65 years of age.
5. Patient has estimated glomerular filtration rate (eGFR) ≥30 mL/min using the Cockcroft-Gault formula.
6. Willing to participate in this study, signed Informed Consent and willing to participate in regular follow-up during the study.
7. Able to understand and cooperate with study procedures. -

Exclusion Criteria:

1. Subjects hospitalized (a) Patients with severe or critical forms of COVID-19 illness or those who are on ventilator support, ECMO, or shock requiring vasopressor support or those with cytokine storm; even not in hospital (b) Patients hospitalized for treatment of severe illnesses (c) "Long COVID-19" syndrome (defined as a diverse set of symptoms that persist after a minimum of 4 weeks from the onset of a diagnosed COVID-19 infection. Common symptoms include respiratory system disorders, nervous system and neurocognitive disorders, mental health disorders, metabolic disorders, cardiovascular disorders, gastrointestinal disorders, malaise, fatigue, musculoskeletal pain, and anemia).
2. Patients with known blood dyscrasia and uric acid kidney stones.
3. Females who are pregnant, breast feeding, or planning a pregnancy.
4. Females of childbearing potential who do not agree to utilize an adequate effective form of contraception.
5. Males with partners of child-bearing potential unwilling to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence effective from the first administration of any of the IPs throughout the trial.

   1. Men with partners of child-bearing potential unwilling to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel, or sexual abstinence. Men with pregnant or lactating partners unwilling to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the fetus or neonate.
   2. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the patients. Periodic abstinence (e.g., calendar, ovulation, sympathothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
6. History of alcohol, chemical, or drug abuse or dependence as per DSM IV criteria within past 6 months.
7. Current active malignancy or history of malignancy within the past five years.
8. Known hypersensitivity history to Investigational Products or any of its component.
9. Any patient on the following medications: Erdafitinib- Lasmiditan- Quinidine due to potential severe drug interaction.
10. Patients with the following conditions:

    1. Immunosuppression
    2. HIV
    3. Current neoplasms
11. Has a history of hepatitis B virus (HBV) or hepatitis C virus (HCV) with cirrhosis, end-stage liver disease, hepatocellular carcinoma.
12. Any other clinically significant abnormal medical condition, which in the Investigator's judgment, would put the patient at increased risk of illness or injury would interfere with study participation or would interfere with the evaluation or quality of the data.
13. Investigator's judgment that participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments including but not limited to: participants who are not expected to survive longer than 48 hours after randomization, or participants with a recent history of mechanical ventilation, or participants with conditions that could limit gastrointestinal absorption of capsule contents.
14. Is taking or is anticipated to require any prohibited medications or therapies.
15. Participation in another trial within previous 3 months and is unwilling to abstain from participating in another interventional clinical study through Day 28 with an investigational compound or device, including those for COVID-19 therapeutics.
16. Any patient that is already taking Investigational Medicinal Products. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Time to Viral Clearance | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: David E Martin, PharmD, Study Director — TrippBio, Inc.
Locations (1):
- PCMCs PGI Yashwantrao Chavan Memorial Hospital, Pune, India

REFERENCES:
- [Derived] Martin DE, Pandey N, Chavda P, Singh G, Sutariya R, Sancilio F, Tripp RA. Oral Probenecid for Nonhospitalized Adults with Symptomatic Mild-to-Moderate COVID-19. Viruses. 2023 Jul 6;15(7):1508. doi: 10.3390/v15071508. PMID 37515194